CLINICAL TRIAL: NCT06004440
Title: A Multi-Center, Prospective, Single-Arm, Observational Study to Evaluate Real-World Outcomes for the Shape-Sensing Ion Endoluminal System
Brief Title: Real World Registry for Use of the Ion Endoluminal System
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: IntuitiveSurgical
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer; Multiple Pulmonary Nodules; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases
Keywords: pulmonary biopsy; pulmonary lesion localization; shape sensing robotic assisted bronchoscopy; ION; Intuitive
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with biopsy, with or without localization, of pulmonary lesion using Ion Endoluminal System: Subjects in which a pulmonary lesion biopsy, with or without localization, was attempted or performed with the Ion Endoluminal System.
  Interventions: Device: Ion Endoluminal System

INTERVENTIONS:
Device: Ion Endoluminal System — Subjects will under a planned procedure with the Ion Endoluminal System

SUMMARY:
The primary objective of this study is to evaluate the performance of the Ion Endoluminal System with real-world use for pulmonary lesion localization or biopsy.

DETAILED DESCRIPTION:
This study is a single-arm, post-market, prospective, multi-center, observational study of subjects undergoing a shape-sensing robotic-assisted bronchoscopy lung lesion localization or biopsy procedure with the Ion Endoluminal System. The primary outcome of this study is focused on evaluating the performance characteristics of the pulmonary lesion biopsy procedure as evaluated by diagnostic yield.

Clinical trial registration is submitted voluntarily under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older at the time of the index procedure.
* Subject is a candidate for an elective, planned lung lesion localization or biopsy procedure utilizing the Ion Endoluminal System.
* Subject able to understand and adhere to study requirements and provide informed consent.

Exclusion Criteria:

* Subject is under the care of a Legally Authorized Representative (LAR) and is unable to provide informed consent on their own accord.
* Subject is participating in an interventional research study or research study investigational agents with an unknown safety profile that would interfere with participation in this study.
* Female subjects who are pregnant or nursing at the time of the index bronchoscopy procedure, as determined by standard site practices.
* Subjects that are incarcerated or institutionalized under court order, or other vulnerable populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled for an elective pulmonary lesion biopsy or localization procedure using the Ion Endoluminal System, 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint to Assess Diagnostic Yield | Intra-procedure through the 24 month follow up period
  Defined as the sum of true positives and true negatives divided by the total number of nodules biopsied. Primary outcome analyses will exclude subjects that are enrolled for localization procedure only.

SECONDARY OUTCOMES:
Secondary Endpoint to Assess Pneumothorax | Intra-procedure through the 30 day follow up period
  Defined as the incidence of subjects that undergo an Ion Procedure with a pneumothorax event, requiring intervention
Secondary Endpoint to Assess Bleeding | Intra-procedure through the 30 day follow up period
  Defined as the incidence of subjects that undergo an Ion Procedure with a bleeding event, with a grade of greater than 2 on the Nashville Scale

CONTACTS AND LOCATIONS:
Overall Officials: Janani Reisenauer, MD, Study Chair — Mayo Clinic; Michael Pritchett, DO, MPH, Study Chair — FirstHealth of the Carolinas
Locations (16):
- United States (16):
  - Orlando Health Orlando Regional Medical Center, Orlando, Florida
  - Ascension Alexian Brothers, Elk Grove Village, Illinois
  - Blessing Hospital, Quincy, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Tulane University, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mercy Hospital of Buffalo, Buffalo, New York
  - Atrium Health of the Carolinas, Charlotte, North Carolina
  - Cone Health Moses Cone Memorial Hospital, Greensboro, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Centennial Medical Center, Nashville, Tennessee
  - Methodist Hospital, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - Aurora Medical Center Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No